CLINICAL TRIAL: NCT00873483
Title: Multicenter, Open-Label, Uncontrolled Study to Investigate the Impact of Weight and BMI on Inhibition of Ovulation of a Transdermal Patch Formulation Containing 0.55 mg Ethinylestradiol and 2.1 mg Gestodene in Young Female Volunteers Stratified by BMI Over a Period of 3 Treatment Cycles
Brief Title: US Ovulation Inhibition Study in Obese Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13871
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Contraception
Keywords: Pregnancy prevention; female contraception; patch
MeSH Terms: interventions — Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — 0.55 mg ethinyl estradiol & 2.1 mg gestodene, 21 days for 3 cycles

SUMMARY:
Birth Control Patch Study

ELIGIBILITY:
Inclusion Criteria:

* Female subject requesting contraception
* Age: 18 - 35 years (inclusive); smokers must not be older than 30 years at the time of informed consent
* Normal cervical smear not requiring further follow-up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the previous 6 months)
* History of regular cyclic menstrual periods
* Willingness to use non-hormonal methods of contraception during the entire study.

Exclusion Criteria:

* Pregnancy or lactation (less than 3 menstrual cycles since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drug
* Significant skin reaction to transdermal preparations or sensitivity to surgical/medical tape
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug (e.g., known skin disease with suspected alteration of dermal absorption or poor adherence of the patch such as psoriasis)
* Any disease or condition that may worsen under hormonal treatment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2010-03-03 (Actual); Study Completion 2010-03-03 (Actual)

PRIMARY OUTCOMES:
Determination of Hoogland Scores | Treatment Cycles 2 & 3

SECONDARY OUTCOMES:
Laboratory values for E2, progesterone, FSH and LH | Pretreatment & regularly during Treatment Cycles 1, 2, 3
Endometrial thickness | Pretreatment & regularly during Treatment Cycles 1, 2, 3
Follicle size | Pretreatment & regularly during Treatment Cycles 1, 2, 3

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- United States (6):
  - Tucson, Arizona
  - San Diego, California
  - Sandy Springs, Georgia
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington